CLINICAL TRIAL: NCT07337525
Title: A Phase 1 Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PLT012 in Patients With Advanced Solid Tumors
Brief Title: A First in Human Study of PLT012 in Participants With Solid Tumor Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pilatus Biosciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLT012-P1-001
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Tumor; Solid Tumor Cancer
Keywords: Gastrointestinal cancer; Liver metastases; Bladder cancer; Liver cancer; Phase 1; Dose escalation; Advanced solid tumors
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urinary Bladder Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm: PLT012 (Experimental): PLT012 administered via intravenous infusion once every 3 weeks
  Interventions: Drug: PLT012

INTERVENTIONS:
Drug: PLT012 — PLT012 (anti-CD36 monoclonal antibody)

SUMMARY:
The goal of this clinical trial is to learn about what doses of PLT012 are safe to use in adults with advanced cancers in solid tumors. It will also learn about how effective different doses of PLT012 are in treating cancer. The main questions it aims to answer are:

What adverse events and toxicities (harmful side effects) are associated with different doses of PLT012? What are the blood levels of PLT012 in your body at different timepoints? What effect does PLT012 have on reducing tumor size and/or preventing the worsening of cancer? All participants will receive PLT012 and none will receive placebo (a look-alike substance that contains no drug).

Participants will receive PLT012 by intravenous infusion once every 3 weeks. Treatment with PLT012 can continue until the participant's disease worsens or they cannot tolerate treatment.

For the first 12 weeks, visits to the clinic will be more frequent (from 1 to 5 times over a 3-week period). After the first 12 weeks, visits will be reduced to once every 3 weeks.

DETAILED DESCRIPTION:
This study is a phase 1, open label, dose escalation study using an initial single participant cohort followed by a BOIN design to evaluate multiple ascending doses of PLT012.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years and provided written informed consent
* Histologically or cytologically confirmed advanced solid tumors (except primary CNS malignancies)
* Has at least one measurable lesion per RECIST v1.1
* ECOG PS of 0 to 1
* Life expectancy of ≥ 12 weeks
* Child-Pugh score of Class A (for hepatocellular carcinoma only)
* Adequate organ function as defined by protocol-specified laboratory values
* Not pregnant or breastfeeding

Exclusion Criteria:

* Insufficient washout period from prior therapies as defined in the study protocol
* Ongoing Grade 2 or higher toxicities from prior treatments (with some exceptions)
* Concurrent or recent (within 2 years) malignancy other than the disease under study (with some exceptions)
* Uncontrolled HIV, uncontrolled hepatitis B, or uncontrolled acute hepatitis C infections
* Unstable/uncontrolled or untreated central nervous system (CNS) metastasis
* Active or recent (within 3 years) autoimmune disease requiring medical treatment
* Recipient of any organ transplant including allogeneic stem-cell transplant
* Clinically significant and active cardiovascular disease
* Known active alcohol or drug abuse
* Psychiatric disorders that would prohibit the understanding of the Informed Consent Form
* Ascites requiring therapeutic paracentesis or hepatic encephalopathy requiring medical interventions within the past 6 months (if hepatocellular carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Frequency, type and severity of dose limiting toxicities and adverse events | 18 months
  Frequency, type and severity of dose limiting toxicities and adverse events according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetic Properties of PLT012 | 18 months
  Plasma concentration of PLT012 at each timepoint at different dose levels
Immunogenicity of PLT012 | 18 months
  Percentage and titer of the anti-drug antibody (ADA) at different dose levels of PLT012
Preliminary efficacy of PLT012 | 18 months
  Clinical activity as evidenced by Overall Response Rate (ORR)
Preliminary efficacy of PLT012 | 18 months
  Clinical activity as evidenced by disease control rate (DCR)
Preliminary efficacy of PLT012 | 18 months
  Clinical activity as evidenced by time to response (TTR)
Preliminary efficacy of PLT012 | 18 months
  Clinical activity as evidenced by duration of response (DOR)
Preliminary efficacy of PLT012 | 18 months
  Clinical activity as evidenced by progression-free survival (PFS)
Preliminary efficacy of PLT012 | 18 months
  Clinical activity as evidenced by overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: Undecided
Pilatus will likely provide this data, but need to formalize the plan first.